CLINICAL TRIAL: NCT01141829
Title: NADPH Oxidase p22phox Polymorphisms and Oxidative Stress in Patients With Obstructive Sleep Apnea
Brief Title: NADPH Oxidase Polymorphisms in Obstructive Sleep Apnea Syndrome (OSAS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Spanish Research Center for Respiratory Diseases (Other)
Responsible Party: Javier Piérola Lopetegui, Hospital Universitario Son Dureta
Other Study IDs: NADPHPM2010
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-01

CONDITIONS: Sleep Apnea Syndrome; Oxidative Stress; Single Nucleotide Polymorphism
Keywords: NADPH oxidase
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Obstructive Sleep Apnea (OSA) is associated with increased oxidative stress. The major sources of Reactive Oxygen Species (ROS) in the vasculature are the NADPH oxidases. Several polymorphisms related to NADPH oxidase expression or NADPH oxidase activity has been identified. The investigators are going to compare the distribution of the allelic frequencies of A-930G and C242T polymorphisms and their possible relationship with the levels of 8-isoprostanes as a marker of oxidative stress in patients with OSA and in a control group without OSA.

DETAILED DESCRIPTION:
DESIGN: CASE-CONTROL STUDY METHODS: We are going to determine the A-930G and C242T p22phox genotypes in patients with OSA and healthy subjects recruited from sleep unit of Son Dureta University Hospital, (Palma de Mallorca, Spain). 8-Isoprostane is going to be measured as an oxidative stress marker with an 8-isoprostane EIA kit (Cayman Chemicals Company, USA) in plasma samples.

ELIGIBILITY:
Inclusion Criteria:Polyysomnografic study with Apnoea/Hypoapnoea Index higher to 10 in patients and lower in controls.

Exclusion Criteria:

* chronic obstructive pulmonary disease, liver cirrhosis, thyroid dysfunction, rheumatoid arthritis, chronic renal failure and/or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with OSAS defined by an apnea hypopnea index (AHI)>10 h-1 will be included in the study along with control subjects without OSAS. Participants were consequently studied at the sleep unit of Hospital Universitario Son Dureta, (Palma de Mallorca, Spain).
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain